CLINICAL TRIAL: NCT04869761
Title: Allogeneic Mesenchymal Stem Cell Therapy in Patients With Chronic Kidney Disease: A Phase I Study
Brief Title: Stem Cell Therapy for Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LaTonya J. Hickson (Other)
Responsible Party: Sponsor-Investigator, LaTonya J. Hickson, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-008380
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Mellitus; Diabetic Nephropathies
Keywords: Stem cell; mesenchymal stem cell; mesenchymal stromal cell; diabetes mellitus; diabetic nephropathy; diabetic kidney disease; kidney; GFR
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Mellitus; Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Arm 1 (Experimental): Subjects with chronic kidney disease will receive allogeneic adipose tissue-derived mesenchymal stem cells (MSC) in two intravenous infusions of 75x10^6 cells at day 0 and month 3.
  Interventions: Drug: Allogeneic adipose-derived mesenchymal stem cells (MSC)-Two Infusions
- Dose Arm 2 (Experimental): Subjects with chronic kidney disease will receive a single intravenous infusion of allogeneic adipose tissue-derived mesenchymal stem cells (MSC) of 150x10^6 cells at day 0.
  Interventions: Drug: Allogeneic adipose-derived mesenchymal stem cells (MSC)-Single Infusion

INTERVENTIONS:
Drug: Allogeneic adipose-derived mesenchymal stem cells (MSC)-Single Infusion — Single MSC infusion of 150x10^6 cells at time zero; intravenous delivery
  Arms: Dose Arm 2
Drug: Allogeneic adipose-derived mesenchymal stem cells (MSC)-Two Infusions — Two MSC infusions of 75x10^6 cells at time zero and three months; intravenous delivery
  Arms: Dose Arm 1

SUMMARY:
The purpose of this study is to assess the safety and tolerability of allogeneic mesenchymal stem / stromal cell therapy in individuals with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years.
* Estimated glomerular filtration rate (eGFR) 25-55 ml/min/1.73m^2
* Spot urine albumin:creatinine ≥30 mg/g unless on Renin-angiotensin-aldosterone system (RAAS) inhibition.
* Ability to give informed consent.

Exclusion Criteria:

* Hemoglobin A1c greater than or equal to 11%.(in individuals with diabetes mellitus)
* Anemia (hemoglobin less than 9g/dL)
* Body weight greater than 150 kg or BMI greater than 50
* Uncontrolled hypertension: sustained systolic blood pressure (SBP) greater than 155 mmHg at screening exam (a maximum of 3 screening visits will be allowed for demonstration of blood pressure control)
* Chronic hypotension: sustained SBP less than 85 mmHg at screening exam.
* Glomerulonephritis not in partial or complete remission for 6 months (or estimated/measured proteinuria greater than 10 grams/day)
* Active glomerulonephritis (glomerular disease) include: ANCA associated glomerulonephritis, post-infectious glomerulonephritis, lupus nephritis, amyloidosis, or other monoclonal gammopathy of renal significance.
* Nephrotic syndrome defined as proteinuria greater than 3.5g per 24 hours, plus hypoalbuminemia (serum albumin less than or equal to 2.5g/L) and edema
* Autosomal dominant or recessive polycystic kidney disease
* Kidney failure requiring renal replacement therapy (hemodialysis, peritoneal dialysis, or kidney transplantation)
* Active immunosuppression therapy (including prednisone greater than or equal to 10mg daily)
* Kidney transplantation history
* Solid organ transplantation history
* Recent cardiovascular event (myocardial infarction, stroke, congestive heart failure) within 6 months or uncontrolled cardiac arrhythmias
* Liver cirrhosis
* Chronic obstructive pulmonary disease, asthma
* History of blood clotting disorder (thromboembolism; pulmonary embolism, deep venous thrombosis)
* Pregnancy
* Active malignancy
* Active infection
* Active hepatitis B or C, or HIV infection
* History of allergic reaction to cellular products (ie. blood transfusions, platelets)
* Active tobacco use
* Illicit drug use and excessive alcohol use presence of psychosocial issues (e.g., uncontrolled mental illness, unpredictable childcare or eldercare responsibilities, irregular/inflexible work schedule) that may interfere with the ability to complete all study procedures
* Subjects anticipating prolonged travel or other physical restrictions that would prohibit return for scheduled study visits
* Inability or unwilling to have magnetic resonance imaging (MRI) or computed tomography (CT) studies
* Inability to give informed consent

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Adverse events and/or serious adverse events | 22 months
  Number of adverse events and/or serious adverse events associated with mesenchymal stem cells intervention

CONTACTS AND LOCATIONS:
Overall Officials: LaTonya Hickson, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel HA, Wang J, Zinn CJ, Learmonth M, Lerman LO, Wolfram J, Hickson LJ. Fortifying the Diabetic Kidney Disease Treatment Armamentarium: Multitarget Senotherapeutic and Regenerative Strategies. J Am Soc Nephrol. 2025 May 7;36(8):1655-1658. doi: 10.1681/ASN.0000000754. No abstract available. PMID 40333016
- [Derived] Andrews TD, Day GS, Irani SR, Kanekiyo T, Hickson LJ. Uremic Toxins, CKD, and Cognitive Dysfunction. J Am Soc Nephrol. 2025 Jun 1;36(6):1208-1226. doi: 10.1681/ASN.0000000675. Epub 2025 Feb 26. PMID 40009460
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials